CLINICAL TRIAL: NCT01122992
Title: Prospective Evaluation of Limbal Relaxing Incision (LRI) in Conjunction With Phacoemulsification Surgery for Astigmatic Correction in Chinese Eyes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Dr Chua Wei Han, Singapore National Eye Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R489/38/2006
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Corneal Astigmatism
Keywords: Limbal relaxing incision; Astigmatic correction; Phacoemulsification surgery; Chinese eyes
MeSH Terms: conditions — Astigmatism

INTERVENTIONS:
Procedure: Limbal relaxing incision

SUMMARY:
The main purpose of this study is to evaluate the use of limbal relaxing incision (LRI) for astigmatic correction. LRI is a procedure where a pair of incisions is made in the peripheral part of the cornea so as to alter its shape and improve the focusing power of the eye.

DETAILED DESCRIPTION:
An important aim in cataract surgery has always been a good postoperative visual outcome. Efforts have been made to achieve this, with the introduction of intraocular lens in the 1980s and small incision cataract surgery in the 1990s. In the recent years, 'refractive' cataract surgery has taken the form of corneal astigmatic correction. Patients with pre-existing astigmatism of more than 1.5D may benefit from surgical correction during cataract surgery, in the hope of improving uncorrected visual acuity as well as lesser image distortion from corneal aberrations.

The limbal relaxing incisional technique involves placement of incisions corresponding to the steep meridian, thereby resulting in corneal flattening and reduction of astigmatic power. It is increasingly popular due to its advantages. LRI is simple to perform, very safe procedure in experienced hands, effective for astigmatic reduction of up to 4D, has rapid visual rehabilitation and is associated with very few visual complications due to the peripheral location of the incisions. Possible complications include globe weakening, corneal perforation, worsening of astigmatism, incorrect incisional placement and corneal hypoesthesia.

LRI technique and the practical nomograms has been described and made feasible by both James P Gills and Louis D Nichamin. Based on preoperatively measured astigmatic power and axis, these two nomograms recommend a systematic approach to the amount of surgical correction required.

The reason for the Nichamin nomogram being more frequently applied, can be attributed to a few inherent features. It accounts for the age of the patient as a surgical variability and recommends the use of paired arcuate limbal incisions measured in degrees of arc. Paired incisions enable symmetric corneal flattening at the steep meridian, whilst arcuate incisions are more physiological, thereby resulting in accurate astigmatic correction that is independent of corneal diameter. Nichamin has also implemented a modified Nichamin age and pachymetry-adjusted nomogram (otherwise known as 'NAPA' nomogram). It accounts for the patient's peripheral corneal thickness and adjusts the incisional depth accordingly to achieve 90% of corneal thickness.

Many studies have shown that LRI is an effective option for astigmatic correction in Caucasian eyes. Whether these results can be further extrapolated to apply to Chinese eyes are still largely uncertain. To date, there has not been a formal study conducted to evaluate this hypothesis. Moreover, there has been some anecdotal evidence suggesting less favorable postoperative outcome of LRI in Chinese eyes. The main objective of our study is thus to assess the utility and effectiveness of LRI in Chinese eyes.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects should be at least 21 years old, and not older than 60 years old
* Only Chinese patients will be eligible for this study
* Presence of a pre-existing regular astigmatism ranging between -1.00 to -3.00D
* Informed consent obtained for both phacoemulsification surgery and LRI procedure
* Study subject is agreeable to comply with the postoperative follow-up regime stated
* Absence of any exclusion criteria

Exclusion Criteria:

* Presence of irregular astigmatism
* Pre-existing pterygium
* Previous corneal / anterior segment surgery
* Pre-existing corneal scar
* Pre-existing corneal pathology eg keratoconus, Fuch's endothelial dystrophy, PUK, etc
* Pre-existing glaucoma

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Amount of surgically induced astigmatism at three months postop | at three months postop

SECONDARY OUTCOMES:
Depth of LRI achieved at one month postop | at one month postop
Unaided visual acuity at three months postop | at three months postop

CONTACTS AND LOCATIONS:
Overall Officials: Wei Han Chua, FRCS Ophthalmology, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Result] Muller-Jensen K, Fischer P, Siepe U. Limbal relaxing incisions to correct astigmatism in clear corneal cataract surgery. J Refract Surg. 1999 Sep-Oct;15(5):586-9. doi: 10.3928/1081-597X-19990901-12. PMID 10504084
- [Result] Gills JP. Treating astigmatism at the time of cataract surgery. Curr Opin Ophthalmol. 2002 Feb;13(1):2-6. doi: 10.1097/00055735-200202000-00002. PMID 11807381
- [Result] Budak K, Friedman NJ, Koch DD. Limbal relaxing incisions with cataract surgery. J Cataract Refract Surg. 1998 Apr;24(4):503-8. doi: 10.1016/s0886-3350(98)80292-7. PMID 9584246